CLINICAL TRIAL: NCT05352100
Title: Testing of a New Therapeutic Vibration Device to Reduce Neuromuscular Weakness in Hospitalized Patients (Hospital Testing)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Researchers decided to move to another technological platform which will require a new record when that research is ready to launch.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Benjamin Bassin, Professor in the Department of Emergency Medicine, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00129402b
Record Dates: First submitted 2022-04-22; First posted 2022-04-28 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Critically Ill
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Hospitalized patients (Experimental): This phase will recruit hospitalized bedridden patients who will be vibrated with the prototype device using various vibration frequencies to determine which frequency produces the optimal physiologic response. Physiologic responses will be determined with a number of devices capable of measuring such things as tissue oxygenation, oxygen consumption, and muscle activity. Blood samples will also be taken to measure certain chemical markers associated with activity and increase blood flow. They may receive multiple 5 minute episodes of various vibration frequencies.
  Interventions: Diagnostic Test: Therapeutic Vibration Device

INTERVENTIONS:
Diagnostic Test: Therapeutic Vibration Device — The Therapeutic Vibration Device is capable of applying force through the axial skeletal spine, through bidirectional compression loading (or prestressing) between the shoulder and the plantar surfaces of the feet. It is placed around the body like a mobile frame so that the applied vibration can affect the whole body. The vibration actuators (drivers) are mobile and can vary in size, frequency response, and force. The design minimizes the possibility of mechanical interference for ventilated/intubated patients.

SUMMARY:
Objective: Test the ability of vibration to produce physiologic, biochemical, and anatomic changes consistent with exercise that would help prevent the development of muscle weakness that occurs when patients are immobile for long periods of time.

DETAILED DESCRIPTION:
During critical illness, patients who are immobilized for more than a few days develop severe muscle and nerve weakness despite receiving full supportive care, which may include physical therapy. In patients requiring mechanical ventilation (a device that breaths for them) for longer than 7 days, the incidence of ICU-acquired weakness is reported to be between 25% and 60%. Such weakness may contribute to increased duration of mechanical ventilation, increased length of stay in the ICU and hospital, and poor quality of life among survivors. This is part of the newly recognized Post Intensive Care Syndrome (PICS). Moreover, patients who are transferred from the ICU to a high-dependency unit (HDU), intensive therapy unit (ITU), post-operative therapy or outpatient ambulatory care need to be mobile as well as awake for any physical therapy. Patients affected by sepsis (severe blood stream infections), osteoarthritis, spinal cord injury, stroke, multiple sclerosis, cerebral palsy, cancer, and other illnesses suffer muscle loss and weakness. Early mobilization (EM) has demonstrated the ability to significantly reduce the detrimental effects of prolonged immobilization such as polyneuropathy and myopathy (nerve damage and muscle weakness), which in turn reduces the time patients spend on mechanical ventilation and the overall length of hospital stay. EM treatments include intense physical therapy, cycle ergometry, transcutaneous electrical muscle stimulation (TEMS) and continuous lateral rotational therapy (CLRT). However, carrying out intense physical therapy using therapists is impractical (especially at smaller hospitals) and cannot be implemented in heavily sedated patients (patients who cannot cooperate). Evidence suggests that vibration may be capable of producing adequate muscle contraction via muscle-spinal loops that may be sufficient to reduce or prevent nerve damage and muscle weakness caused by prolonged immobilization thus serving as an effective treatment making patients stronger when they leave the ICU.

The purpose of this study is to test a prototype vibration device and strategy on its ability to exercise large muscle groups, increase muscle blood flow, and increase circulating levels of blood chemicals associated with exercise/activity. The study will be used to find optimal vibration frequencies that provide maximal evidence of associated muscle activity. Eventually the investigators hope to see a vibration device capable of delivering a more effective therapy compared to the smaller gains derived from traditional measures of physical therapy in critically ill patients such as TEMS, CLRT and cycle ergometry to patients. The vibration device may directly benefit the patient in terms of health, length of stay and reduced re-admission, hospital staff in terms of productivity (i.e., through reduction in nursing effort) and the hospital in terms of reduced cost and return on investment. Its value is also envisioned in many other populations of immobilized acutely ill and injured patients as well as those with chronic conditions.

Originally registered as a single record, (NCT03479008) this registration represents the intervention and outcomes of testing with hospitalized patients. NCT03479008 will remain open until it is certain that no additional modifications of the device are required to go through a new round of iterative testing with healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* sick patients admitted to the ICUs at University of Michigan hospital

Exclusion Criteria:

1. Acute Spinal Cord Injury
2. Acute vertebral body fracture or injury
3. Acute stroke or intracerebral hemorrhage
4. Hemodynamic instability or other event/condition believed by care team to warrant nonparticipation
5. Known pregnancy
6. Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-11 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
StO2 | 2 hours
  Tissue hemoglobin oxygen saturation (StO2) using near infrared spectroscopy of the thighs, biceps, and brain.
VO2 | 2 hours
  Oxygen consumption using a VO2 monitor and mask
EMG | 2 hours
  Muscle contraction using noninvasive electromyography
Blood markers - serum glucose | On the day of device use (1 day)
  Serum glucose (mg/dl)
Blood markers - lipids | On the day of device use (1 day)
  lipids (mg/dl)
Blood markers - cytokines | On the day of device use (1 day)
  inflammatory cytokines IL-6, TNFα, IL-1β (pg/ml)
Blood markers - growth hormone | On the day of device use (1 day)
  growth hormone (ng/ml)
Blood markers - cortisol | On the day of device use (1 day)
  cortisol (μg/dL)
bone turnover markers | On the day of device use (1 day)
  C-terminal telopeptide of type I collagen (CTX-I) and tartrate-resistant acid phosphatase 5b (U/L)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin S Bassin, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No